CLINICAL TRIAL: NCT05485857
Title: Influence of Arrangement of Small Intestine Order on the Recovery of Bowel Function After Laparoscopic Colorectal Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Head of colorectal surgery, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHCS-intestine
Record Dates: First submitted 2022-07-24; First posted 2022-08-03 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arrangement group (Experimental): Experimental group: After the completion of laparoscopic-assisted colorectal cancer surgery, the chief surgeon performed laparoscopic small bowel arrangement before closing the abdomen, straightening the small bowel from the colon-small bowel anastomosis or the ileocecal valve to the ligament of Trevor, and restoring the original position of the small bowel. Afterwards, close the abdomen.
  Interventions: Procedure: Arrangement of small intestine order before close the abdomen
- No arrangement group (No Intervention): No arrangement group: After completing the routine operation of laparoscopic-assisted colorectal cancer surgery, the abdomen was closed directly.

INTERVENTIONS:
Procedure: Arrangement of small intestine order before close the abdomen — After the completion of laparoscopic-assisted colorectal cancer surgery, the chief surgeon performed laparoscopic small bowel arrangement before closing the abdomen, straightening the small bowel from the colon-small bowel anastomosis or the ileocecal valve to the ligament of Trevor, and restoring the original position of the small bowel. Afterward, close the abdomen.
  Arms: Arrangement group

SUMMARY:
The method of arranging and restoring the position of the small intestine under laparoscopy is used to determine whether it can promote the recovery of intestinal function after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed colorectal cancer, patients undergoing colon cancer or radical resection of high rectal cancer；
* Tumor Stage (TNM): I-III；
* Age: >18 years old; <80 years old;
* ASA: I-III;
* Agree and sign the informed consent form.

Exclusion Criteria:

* Stoma patients；
* Patients with preoperative intestinal obstruction；
* Constipation patients (More than three days before the last bowel movement)；
* Combined other organ resection patients；
* Stroke or spinal cord injury patients；
* Long-term opioid use patients；
* Patients with a history of previous abdominal surgery；
* Patients refused entry into the trial；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
First flatus time after surgery | 50 hours
  The investigators will record the time from the end of the surgery to the patient's first flatus time by hours.

SECONDARY OUTCOMES:
Time to liquid diet | 70 hours
  The investigators will record the time from the end of the surgery to the patient's first diet time by hours.
Postoperative hospital stay | 30 days
  The investigators will record the time from the end of the surgery to the patient's decharge time by days.
Paralytic ileus time after surgery | 30 days
  The investigators will record the time after surgery if the patient's first fluid time is more than seven days after the operation.
First defecate time after surgery | 70 hours
  The investigators will record the time from the end of the surgery to the patient's first defecate time by hours.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No